CLINICAL TRIAL: NCT02752243
Title: A Prospective Phase I/II Study to Investigate the Feasibility, Safety and Efficacy of IL-15 Activated Cytokine Induced Killer (CIK) Cells in Relapsing Patients With Acute Leukemia or Myelodysplastic Syndromes After Allogeneic SCT
Brief Title: CIK-Cells in Relapsing Patients With Acute Leukemia or Myelodysplastic Syndromes After SCT.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peter Bader (Other)
Responsible Party: Sponsor-Investigator, Peter Bader, Prof. Dr. med., Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFM-CIK-Cell Study 01; 2013-005446-11 (EudraCT Number)
Record Dates: First submitted 2016-03-31; First posted 2016-04-26 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Myelodysplastic Syndromes; Acute Leukemia
Keywords: acute leukemia; myelodysplastic syndrome (MDS); Stem Cell Transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CIK-Cells (Experimental): IL-15 activated CIK cells individually generated from PB mononuclear cells of the original stem cell donors.
  Interventions: Drug: CIK-Cells

INTERVENTIONS:
Drug: CIK-Cells — IL-15 activated CIK cells individually generated from PB mononuclear cells of the original stem cell donors.

SUMMARY:
Multi-site, non-randomized Phase I/II study involving children and adults.

DETAILED DESCRIPTION:
This is a phase I/II multicenter-study to investigate the feasibility safety and efficacy of interleukin (IL)-15 activated CIK cells in patients with acute leukemia or myelodysplastic syndrome (MDS) showing evidence of relapse after allogeneic stem cell transplantation (SCT).

CIK cell infusions will be given with an interval of 4-6 weeks according to a dose escalation schedule in patients with impending relapse after allogeneic SCT. In presence of acute graft versus host disease (aGvHD) ≥ grade II, the next scheduled infusion will not be administered.

ELIGIBILITY:
Inclusion Criteria:

Acute leukemia and MDS patients with molecular or cytogenetic relapse in peripheral blood (PB) or bone marrow (BM) samples obtained during monitoring for relapse after allogeneic SCT.

MRD detected by Ig/TCR gene rearrangement testing or any detected disease specific DNA or RNA sequence or disease specific cell surface Proteins or mixed recipient chimerism (MC) ≥ 1% and < 40%, or levels ≥ 10-4 of BCR-ABL/ABL ratio or any other disease specific cytogenetic abnormality will trigger CIK cell interventions.

* Respecting MC, MC = 1% of autologous/recipient signals in PB samples must be confirmed by another PB or BM sample within one week. Patients with MC = 1% of autologous/recipient signals in CD33+ and/or CD34+ subpopulations in PB samples must be confirmed by BM analyses within one week. Acute leukemia and MDS patients with MC = 1% of autologous/recipient signals including signals in CD33+ and/or CD34+ subpopulations in BM samples must not be confirmed.
* Acute leukemia and MDS patients with frank relapse ≥ 120 days after allogeneic SCT who achieved complete remission (CR) or blast clearance (i.e. <5% blasts) in the bone marrow after re-induction chemotherapy.
* All patients must be in complete remission or have achieved blast clearance (i.e. <5% blasts) in the bone marrow before 1st CIK cell treatment (bone marrow assessment at a maximum of 7 days in advance of 1st treatment is obligatory).
* Patients without immunosuppressive agents and steroids for at least 7 days.
* Patients without chemo- or immune therapy during CIK cell treatment, except patients with thyrosine-kinase inhibitors (TKI) for treatment of BCR-ABL positive leukemia. Last DLI treatment must be 4 weeks before 1st CIK cell treatment.
* Patients with < grade II aGvHD.
* Patients with Karnowsky or Lansky performance status ≥ 50%.
* Patients and/or his/her legal representative having reviewed the patient information/informed consent form and have had their questions answered and have given written informed consent.

Exclusion Criteria:

* Acute leukemia and MDS patients with hematologic relapse < day 120 after allogeneic stem cell transplantation.
* Patients with 5% and more malignant cells in a representative bone marrow analysis performed at a maximum of 7 days before 1st CIK cell treatment (obligatory).
* Patients with immunosuppressive agents or steroids.
* Patients with chemo- or immune therapy, except patients with thyrosine-kinase inhibitors (TKI) for BCR-ABL positive leukemias.
* Patients with ≥ grade II GvHD.
* Patients with rapid T cell regeneration and any signs of GvHD
* Patients with Karnowsky or Lansky performance status < 50%.
* Patients and/or his/her legal representative having reviewed the patient information/informed consent form and have had their questions answered and have not given written informed consent.
* HIV-positive patients.
* HBV/HCV positive patients.
* Patients with prior solid organ transplantation.
* Patients treated with any other investigational product within the last 28 days or five half-lives (whichever is longer).
* Hypersensitivity to any component of the study drug
* Female patients of child-bearing potential not agreeing to use a highly effective method of birth control resulting in a low failure rate (i.e. < 1%) when used consistently and correctly.
* Male patients with female partners of childbearing potential not agreeing to use a highly effective method birth control resulting in a low failure rate (i.e. < 1%) when used consistently and correctly.
* Pregnancy/Breastfeeding.
* Patients with severe infections or signs/symptoms of infection within 2 weeks prior to study start.

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-03; Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The occurrence of grade three or four acute Graft versus Host Disease (aGvHD) | two until four weeks after CIK-Cell Infusion
Extensive chronic Graft versus Host Disease (cGvHD) | two until four weeks after CIK-Cell Infusion

SECONDARY OUTCOMES:
Efficacy of CIK-Cells analyzed by progression free survival | one year
Overall survival | one year

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - University Hospital Heidelberg, Ruprecht Karls University, Hospital for children and adolescents, Pediatrics III, Department of Oncology, Haematology, Immunology and Pneumology, Heidelberg, Baden-Wurttemberg
  - Division for Stem Cell Transplantation and Immunology, Department for Children and Adolescents, University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Internal Medicine II, Department of Hematology, Oncology, Rheumatology and Infectious Diseases, Goethe-University Frankfurt/Main, Frankfurt am Main, Hesse
  - University Medicine Duesseldorf, Department of Paediatric Oncology, Haematology and Immunology, Bone Marrow Transplantation Unit, Düsseldorf, North Rhine-Westphalia
  - Internal Medicine III, Department of Hematology and Oncology, Johannes Gutenberg University, Mainz, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: No